CLINICAL TRIAL: NCT03563274
Title: Observational, Multicenter Study to Further Confirm The Efficacy and Safety of QuiremSpheres® (Holmium-166 Microspheres) Selective Internal Radiation Therapy (SIRT) in Unresectable Liver Cancer Patients.
Brief Title: QuiremSpheres Observational Study
Acronym: Hope166
Status: Terminated | Type: Observational
Why Stopped: did not meet planned recruitment expectations with a slow recruitment rate
Sponsor: Terumo Europe N.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: T131E1
Record Dates: First submitted 2018-06-08; First posted 2018-06-20 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Liver, Cancer of, Non-Resectable
Keywords: Hepatocellular Carcinoma,Holmium-166,SIRT,QuiremSpheres®
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Selective Internal Radiation Therapy with QuiremSpheres® — The main purpose of this study is to further assess treatment efficacy and safety after using QuiremSpheres® for the treatment of patients with unresectable primary liver cancer or unresectable liver metastases suitable for SIRT and allocated to this treatment by a multidisciplinary tumor board.
  Other Names: SIRT, Radioembolization

SUMMARY:
The main purpose of this study is to further assess treatment efficacy and safety after using QuiremSpheres® for the treatment of patients with unresectable primary liver cancer or unresectable liver metastases suitable for SIRT and allocated to this treatment by a multidisciplinary tumor board.

DETAILED DESCRIPTION:
Liver tumors can be of primary (Hepatocellular Carcinoma, HCC) or metastatic (mainly from colorectal carcinoma, CRC) origin. Both HCC and CRC are common causes of death from cancer worldwide. The overall incidence of HCC and CRC remains high in developing countries and is steadily rising in most industrialized countries. Available treatment options depend on the size, number, and location of tumors, on liver status, overall performance status and comorbidities, on patency of portal vein and presence of extrahepatic metastatic disease. They include surgical (liver resection, liver transplantation), systemic (e.g. chemotherapy, immunotherapy), ablative (thermal ablation, chemical ablation) and intra-arterial (chemoembolization, radioembolization) modalities. Radioembolization, also known as Selective Internal Radiation Therapy (SIRT) with microspheres containing a radiation-emitting isotope (Yttrium-90 or Holmium-166) delivers localized radiation in the vasculature around liver tumors with relatively limited concurrent injury to the surrounding normal/healthy tissue. Yttrium-90 radioembolization is currently included in several guidelines (EASLEORTC, ESMO).

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnosis of primary liver tumor or metastases in the liver from other primary cancers, allocated to SIRT with QuiremSpheres® as decided by a multidisciplinary tumor board
* Patient is ≥ 18 years
* Patient has understood and signed written informed consent to data collection in the study

Exclusion Criteria:

* Patient's refusal
* Local practice guidelines prohibiting the patient to receive SIRT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable primary liver cancer or unresectable metastases in the liver.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Tumor response | 3 months
  1. Tumor response in the liver
  • Tumor response in liver for overall population and each tumor type, assessed 3 months after SIRT has been completed as per routine practice following the corresponding guidelines for each tumor type (e.g. RECIST, mRECIST, EASL)
Safety | 12 months
  2. Frequency and Severity of Adverse Events
  • Safety will be evaluated by monitoring and recording the grade 3, 4 and 5 adverse events (AE) and all adverse device effects (ADE) occurring during and after treatment throughout follow up of patients. Severity of adverse events will be rated following the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Safety assessment will also be based on routine blood tests with an emphasis on the liver function parameters obtained at baseline, after the SIRT procedure and throughout the follow up period.

SECONDARY OUTCOMES:
Time to progression in liver and overall | 12 months
  Time from SIRT procedure until progression in liver / overall progression
Progression free survival in liver and overall | 12 months
  Time from SIRT procedure until progression in liver / overall progression or death.
Overall survival rate | 12 months
  Time from SIRT procedure until death from any cause
Percentage of patients downstaged to surgery, transplantation or any local ablative therapy (RFA/MWA…) | 12 months
  Number of patients that after the SIRT procedure underwent a surgery or transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Dragica Paunovic, MD, Study Director — Chief Medical Officer at Terumo Europe
Locations (2):
- Universitätsklinikum Carl Gustav Carus, Dresden, Germany
- UMC Utrecht, Utrecht, Netherlands